CLINICAL TRIAL: NCT05080374
Title: Effects of Combining High Speed Low Amplitude Spinal Manipulation (HVLA) With Functional Elastic Bandage, Diaphragm Training and a Lumbar Exercise Program in Patients With Nonspecific Low Back Pain: a Randomized Clinical Trial.
Brief Title: Effects of Spinal Manipulation in Patients With Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ignacio Alejandro Astudillo Ganora (Other)
Responsible Party: Sponsor-Investigator, Ignacio Alejandro Astudillo Ganora, Physiotherapist, Phd, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3500/2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Back Pain; Lumbar Pain Syndrome; Back Pain, Low
MeSH Terms: conditions — Back Pain; Somatoform Disorders; Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HVLA + exercise Group (Experimental): Spinal manipulation (HVLA) + trunk exercise program
  Interventions: Other: Spinal Manipulation + exercise program
- HVLA + kinesiotaping group (Experimental): Spinal manipulation (HVLA) + Kinesiotaping (lumbar)
  Interventions: Other: Spinal manipulation + Kinesiotaping
- HVLA + Respiratory exercise group (Experimental): Spinal manipulation (HVLA) + respiratory exercise program
  Interventions: Other: spinal manipulation + respiratory exercise

INTERVENTIONS:
Other: Spinal Manipulation + exercise program — high-speed, low-amplitude spinal manipulation plus a trunk exercise program
  Arms: HVLA + exercise Group
Other: Spinal manipulation + Kinesiotaping — high-speed, low-amplitude spinal manipulation plus elastic bandage (Kinesiotaping) application to the trunk area
  Arms: HVLA + kinesiotaping group
Other: spinal manipulation + respiratory exercise — high-speed, low-amplitude spinal manipulation plus a breathing exercise program for the diaphragmatic muscles
  Arms: HVLA + Respiratory exercise group

SUMMARY:
Introduction: Nonspecific low back pain is the most common cause of visits to medical personnel and is the largest cause of absenteeism in the world. (1), Nonspecific low back pain accounts for 85% of low back pain, notably affecting quality of life and working life (2), There is a 50-70% probability that a person will have low back pain during their life ( 3), lumbago produces 300,000 years lived with disability (ADL), being the first burden of disease in Chile, surpassing hypertensive heart disease and depression (4). There are many therapeutic approaches to the management of nonspecific low back pain, including high-speed, low-amplitude spinal manipulations (5). This technique consists of applying a short and rapid force at the level of the joint that is restricted, in order to restore normal joint mobility. The physiological effects of manipulations are not sufficiently studied, but some authors (6) (7) suggest that the nervous system is the mediator of the effects of spinal manipulation. Among non-pharmacological interventions, numerous clinical guidelines recommend the use of therapeutic exercise for low back pain (8), including a wide variety of types of recommended exercises, the most traditionally recommended being aerobic exercises, exercises that involve stretching postures of the back. vertebral musculature, strengthening and strength exercises (9) and central stabilization exercises (10). Recently, the effects of inspiratory muscle and diaphragm training exercises in patients with low back pain are being investigated (11). The application of an elastic bandage (12) in the lumbar area generates a proprioceptive signal through the skin, producing analgesia and a feeling of support in the area.

Objectives: To compare the effects of different therapeutic approaches in combination with spinal manipulation.

Design and method: Single-blind randomized clinical trial Results: Significant differences are expected before and after treatment and differences between groups.

Conclusion: The aims of this study is to demonstrate that High speed and low amplitude spinal manipulation plus other conservative treatment is a valid therapeutic strategy for the management of nonspecific low back pain

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* with nonspecific low back pain

Exclusion Criteria:

* chronic low back pain (more than 3 months)
* spinal surgeries
* red flags for spinal manipulation (osteoporosis, bone metastasis, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
changes in pain EVA | baseline after 6 weeks and a month
  observe changes in pain through visual analogue scale (VAS) 0 to 10
Changes in pain pressure algometers | baseline after 6 weeks and a month
  observe changes in pain in painful points through a pressure monitor (painmeter) (0 to 10 kilograms 0 to 22 pounds)
Biomechanical changes (lateral tilt test) | baseline after 6 weeks and a month
  observe the changes in the biomechanics of the spine through the lateral tilt test (centimeters from the tip of the middle finger to the ground)
biomechanical changes (finger-floor test) | baseline after 6 weeks and a month
  observe the changes in the biomechanics of the spine through the finger-floor test (centimeters from the tip of the middle finger to the ground)
Biomechanical changes (shober test) | baseline after 6 weeks and a month
  observe the changes in the biomechanics of the spine through the Shober test (Schöber test. It is performed with the patient standing and the examiner on his back. A point is indicated that locates L5 (at the height of the dimples of Venus or the iliac crests are used, which correspond to L4, and is marked 1cm below) and a second point is marked 10cm above.)
changes in function | baseline after 6 weeks and a month
  observe changes in disability due to nonspecific low back pain through the Oswestry test (The Oswestry Test comprises 10 items, of 10 points each, with a maximum of 100, this score being the worst possible functional state.)

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotherapy deparment, Murcia University, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No